CLINICAL TRIAL: NCT07324902
Title: The Effect of Lipoprotein (a) on Arterial Stiffness, Endothelial Function and Left Atrial and Left Ventricular Deformation - An Observational Study.
Brief Title: The Effect of Lipoprotein (a) on Arterial Stiffness, Endothelial Function and Myocardial Deformation
Acronym: Lpa_endo
Status: Recruiting | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Professor of Cardiology, University of Athens
Other Study IDs: 787/01-11-2024
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Lipoprotein Disorder; Arterial Stiffness; Endothelial Dysfunction
Keywords: lipoprotein a; artrial stiffness; endothelial glycocalyx; myocardial deformation; oxidative stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Participants with elevated Lipoprotein a: Group A: PArticipants with elevated Lp(a) (Lp(a) ≥50 mg/dL) with normal Total Cholesterol levels (Cholesterol<200 mg/dl). All participants (n≥100) will undergo assessment of arterial stiffness by measing PWV, evaluation of thickness of endothelial glycocalyx bymeasuring PBR, assessment of myocardial deformation by measuring LA strain and LV GLS and quantification of oxidative stress burden by measuring MDa and PCs at baseline, at 6 months and at 12 months.
- Participants with elevated Total Cholesterol: Group B: PArticipants with normal Lp(a) (Lp(a) <50 mg/dL) with elevated Total Cholesterol levels (Cholesterol ≥200 mg/dl).
  All participants (n≥100) will undergo assessment of arterial stiffness by measing PWV, evaluation of thickness of endothelial glycocalyx bymeasuring PBR, assessment of myocardial deformation by measuring LA strain and LV GLS and quantification of oxidative stress burden by measuring MDa and PCs at baseline, at 6 months and at 12 months.
- Participants with normal lipids levels: Group C: PArticipants with Lp(a) (Lp(a) <50 mg/dL) and TotalCholesterol levels (Cholesterol ≥200 mg/dl) within reference range.
  All participants (n≥100) will undergo assessment of arterial stiffness by measing PWV, evaluation of thickness of endothelial glycocalyx bymeasuring PBR, assessment of myocardial deformation by measuring LA strain and LV GLS and quantification of oxidative stress burden by measuring MDa and PCs at baseline, at 6 months and at 12 months.

SUMMARY:
1. Introduction Lipoprotein(a), or Lp(a), is a type of lipoprotein that is structurally similar to LDL (low-density lipoprotein) but carries an additional protein called apolipoprotein (a).
2. Purpose of the Study

   The primary purpose of this study is to investigate the effect of Lp(a) levels on arterial stiffness, endothelial function, and left atrial (LA) and left ventricular (LV) deformation over a 12-month follow-up period.

   Secondarily, the study will investigate:
   * a) The incidence of major adverse cardiovascular events (MACE), including cardiovascular death, acute myocardial infarction, and acute stroke.
   * b) The correlation between MACE incidence and parameters of arterial stiffness, endothelial function, and LA/LV deformation.
   * c) The levels of oxidative load markers.
3. Materials and Methods This observational study will include adults aged 18-75 years (regardless of gender) who visit the outpatient clinics of the 2nd University Cardiology Clinic at "Attikon" General Hospital. All participants will sign a consent form. A full medical history, clinical examination, and blood collection will be performed to determine levels of Total Cholesterol, LDL-C, HDL-C, triglycerides, and Lp(a) at each visit..

Participants will be divided into three groups:

* Group A: Lp(a) ≥50 mg/dL with Total Cholesterol<200 mg/dl
* Group B : Lp(a) <50 mg/dL. with Total Cholesterol>200 mg/dl
* Group C (Control): Lp(a) <50 mg/dL. with Total Cholesterol<200 mg/dl At each group n ≥ 100 participants are anticipated.

Measurements at baseline, at 6 and at 12 months:

* Arterial Stiffness: Determination of carotid-femoral pulse wave velocity (cf-PWV) using the Complior SP device and 24-hour pulse wave analysis with the Mobil-O-Graph device.
* Endothelial Function: Measurement of the endothelial glycocalyx thickness of sublingual capillaries using a Sidestream Dark Field (SDF) camera (GlycoCheck). This is expressed through the perfused boundary region (PBR) index.
* Cardiac Deformation: Use of two-dimensional strain (speckle tracking) to calculate the Global Longitudinal Strain (GLS) of the LV and LA strain.
* Oxidative Load: Determination of malondialdehyde (MDA) and protein carbonyls (PCs) levels as markers of oxidative stress using spectrophotometric kits.

Statistical Analysis: Comparisons regarding the changes in these markers over 6 and 12 months will be conducted between the three groups.

DETAILED DESCRIPTION:
1. Introduction Lipoprotein(a), or Lp(a), is a type of lipoprotein that is structurally similar to LDL (low-density lipoprotein) but carries an additional protein called apolipoprotein (a). Recent data establishes Lp(a) as a predisposing risk factor for cardiovascular diseases, such as coronary artery disease, stroke, and aortic valve stenosis. Elevated levels of Lp(a) contribute to these conditions by promoting atherosclerosis. Its levels are primarily determined genetically, with minimal influence from diet and lifestyle. This makes it a significant factor for assessing cardiovascular risk, particularly in individuals with a family history of coronary artery disease or patients who experience early cardiovascular problems despite having normal lipid levels.

   While Lp(a) levels can vary greatly, the generally accepted threshold for increased cardiovascular risk is 50 mg/dL (or 125 nmol/L). Individuals with levels above this limit are at a higher risk for cardiovascular events. It is estimated that 20-30% of the general population has elevated Lp(a) levels, making it a common risk factor. Currently, there are no widely available treatments specifically targeting Lp(a) levels, though PCSK9 inhibitors and inclisiran have shown promising results in clinical trials.
2. Purpose of the Study There is currently insufficient bibliographic documentation regarding the effect of Lp(a) on arterial stiffness, endothelial function, and the deformation of the left atrium and left ventricle.

   The primary purpose of this study is to investigate the effect of Lp(a) levels on arterial stiffness, endothelial function, and left atrial (LA) and left ventricular (LV) deformation over a 6-month follow-up period.

   Secondarily, the study will investigate:
   * a) The incidence of major adverse cardiovascular events (MACE), including cardiovascular death, acute myocardial infarction, and acute stroke.
   * b) The correlation between MACE incidence and parameters of arterial stiffness, endothelial function, and LA/LV deformation.
   * c) The levels of oxidative load markers.
3. Materials and Methods

This observational study will include adults aged 18-75 years (regardless of gender) who visit the outpatient clinics of the 2nd University Cardiology Clinic at "Attikon" General Hospital. All participants will sign a consent form. A full medical history, clinical examination, and blood collection will be performed to determine levels of Total Cholesterol, LDL-C, HDL-C, triglycerides, and Lp(a) at each visit. Participants will be divided into three groups:

* Group A: Lp(a) ≥50 mg/dL with Total Cholesterol<200 mg/dl
* Group B : Lp(a) <50 mg/dL. with Total Cholesterol>200 mg/dl
* Group C (Control): Lp(a) <50 mg/dL. with Total Cholesterol<200 mg/dl The exclusion criteria encompass: 1. History of autoimmune/autoinflammatory disease, 2. Severe valvular heart disease, 3. severe chronic kidney disease(eGFR<60 ml/min/1.73 m2), 4. Active Pregnancy and 5. Severe hepatic impairment.

At each group n ≥ 100 participants are anticipated.

The following measurements will be conducted for each group at baseline and after 6 and 12 months post enrollment:

* Arterial Stiffness: Determination of carotid-femoral pulse wave velocity (cf-PWV) using the Complior SP device and 24-hour pulse wave analysis with the Mobil-O-Graph device. Pulse wave velocity is the gold standard for the evaluation of arterial stiffness [21,22]. The investigators will use two non-invasive pressure sensors to record the carotid and femoral waveforms. The investigators will measure the distance between the two arterial sites with a tape measure. PWV is calculated by dividing the distance by transit time between waves (m/s). The appropriate corrections of the PWV were applied, after multiplying the default PWV output values by 0.8 [22]. Central systolic blood pressure (cSBP, mmHg) and central diastolic blood pressure (cDBP, mm Hg) will be measured using Complior.
* Endothelial Function: The investigators will measure the perfused boundary region (PBR) of the sublingual arterial microvessels (ranged from 4 to 25μm) using Sidestream Darkfield (SDF) imaging (Microscan, Glycocheck, Microvascular Health Solutions Inc., Salt Lake City, Utah, United States) [18]. This technique enables the assessment of the endothelial glycocalyx, using a non-invasive method. The PBR is the cell poor layer, which results from the phase separation between the flowing RBC's and plasma on the surface of the microvessel lumen. The PBR includes the most luminal part of glycocalyx that does allow cell penetration. Thus, an increased PBR is consistent with deeper penetration of erythrocytes into glycocalyx, indicating a loss of glycocalyx barrier properties and is a marker of reduced glycocalyx thickness. The measurement of endothelial glycocalyx thickness using SDF imaging is easy to perform (duration of 3 minutes) and is not biased by operator skills. Moreover, it has a standardized methodology, provides measurements of multiple sample sites (>3,000 vascular segments of sublingual microvasculature), has very good reproducibility and thus is proposed as a valid method to assess endothelial integrity by the European Society of Cardiology Working Group on Peripheral Circulation. The PBR measurements are independent of RBC filling of the vessels segments (hematocrit), because the software only includes vessel segments that have a filling percentage more than 50% [9,18]. Hence, vessel segments are only selected when at least 11 of the 21-line markers have a positive signal for the presence of an erythrocyte. Thus, PBR values are independent of hematocrit, reflecting a damaged glycocalyx that is more accessible for circulating erythrocytes.
* Cardiac Deformation: In all participants the investigators will measure longitudinal systolic strain from standard two dimensional (2D) acquisitions (frame rate: 70-80/second) with the use of a dedicated software (EchoPac 206, GE Healthcare). Global longitudinal strain (GLS) is calculated using the 17 LV segment model imaged from apical chamber views (4,2 and 3 chamber view). The myocardial deformations at the basal, mid-ventricular, and apical segments were averaged to GLS. All variables represent the mean value measurements taken in three consecutive cardiac cycles. Inter- and intra- observer variability of GLS was 8 and 5%, respectively. LA function will be evaluated using transthoracic echocardiographic speckle -tracking strain imaging. A speckle -tracking algorithm was applied to the LA myocardium in apical 4- and 2- chamber views. The region of interest width was adjusted to the thickness of the LA wall, and the cardiac cycle was demarcated by indicating QRS onset. LA reservoir strain, a metric of LA compliance, was measured as peak longitudinal strain (average of all 12 segments in the apical 4- and 2- chamber views) during ventricular systole, taking the QRS onset as the reference point. After having defined by anatomical M-mode mitral and aortic valve opening and closure as well as atrial contraction, LA longitudinal strain, obtained by 2D strain, will be measured in all three atrial phases (reservoir, conduit, and atrial contraction) as follows : reservoir period was defined as the interval between mitral valve closure and mitral valve opening, conduit period as the interval between mitral valve opening and the onset of atrial contraction, as assessed by anatomical M- mode, and contractile period as the interval between the onset of atrial contraction, as assessed by anatomical M-mode, and mitral valve closure. Subsequently, the atrial deformation of each period was calculated by measuring the respective difference of strain (values at the end minus values at the beginning).
* Oxidative Load: Determination of malondialdehyde (MDA) and protein carbonyls (PCs) levels as markers of oxidative stress. MDA will be estimated spectrophotometrically with a commercial kit (Oxford Biomedical Research, Rochester Hills, MI) of colorimetric assay for lipid peroxidation (measurements range, 1-20 nmol/l). For the determination of PCs (nmol/mL), the investigators used the spectrophotometric assessment of 2,4-dinitrophenylhydrazine derivatives of PCs.
* Statistical Analysis: Statistical analysis will be conducted by employing SPSS version 29 (IBM SPSS Statistics, Inc., Chicago, IL). All continuous variables variables will be presented as mean ±SD if they are distributed normally, as indicated by the Kolmogorov-Smirnov and Shapiro-Wilk normality tests. In case of non-normal distribution, transformation into ranks will be performed. Nominal variables are presented as percentages. Correlation analysis will be performed via Spearman or Pearson correlation tests, based upon data distribution. Categorical variables are analyzed via either Chi-square tests or Fisher's exact tests, as appropriate. ANOVA for repeated measurements will be used for (1) measurements of the aforementioned at the beginning, at 6 and at 12 months (which is considered a within-subject factor) and (2) also the differenced of different groups, as a between-subject factor). Post-hoc comparisons will be conducted with Bonferroni's correction. The F and the respective P values between the different time periods of measurements will be calculated. Furthermore the F and P values between time of measurement of the biomarkers and the examined groups will be estimated. The Greenhouse-Geisser, Huynh-Feldt or Lower-Bound corrections will be used when the sphericity assumption, as evaluated by Mauchly's test, will not be met. The percent changes of the examined variables after intervention will also be compared by one way ANOVA. All statistical tests are two-tailed and a p-value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adults participants 18-75 years old
* Willing to sign the informed consent and paerticipate in the study

Exclusion Criteria:

* History of autoimmune/autoinflammatory disease,
* Severe valvular heart disease,
* severe chronic kidney disease(eGFR<60 ml/min/1.73 m2),
* Active Pregnancy
* Severe hepatic impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This observational study will include adults aged 18-75 years (regardless of gender) who visit the outpatient clinics of the 2nd University Cardiology Clinic at "Attikon" General Hospital. All participants will sign a consent form. A full medical history, clinical examination, and blood collection will be performed to determine levels of Total Cholesterol, LDL-C, HDL-C, triglycerides, and Lp(a) at each visit. Participants will be divided into three groups:
  * Group A: Lp(a) ≥50 mg/dL with Total Cholesterol<200 mg/dl
  * Group B : Lp(a) <50 mg/dL. with Total Cholesterol>200 mg/dl
  * Group C (Control): Lp(a) <50 mg/dL. with Total Cholesterol<200 mg/dl At each group n ≥ 100 participants are anticipated.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-08-17 (Estimated)

PRIMARY OUTCOMES:
Comparison of endothelial glycocalyx thickness difference between groups | 12 months
  Comparison of Perfused Boundary Region (PBR) difference of sublingual vessels between groups
Comparison of arterial stiffness difference between groups | 12 months
  Comparison of carotid-to-femoral Pulse Wave Velocity (PWV) difference between groups
Comparison of left atrial deformation difference between groups | 12 months
  Comparison of left atrial strain difference between groups
Comparison of left ventricular deformation difference between groups | 12 months
  Comparison of left ventricular strain difference between groups

SECONDARY OUTCOMES:
Comparison of oxidative stress burden difference between groups | 12 monnths
  Comparison of malondialdehyde difference between groups
Comparison of major adverse cardiovascular events between groups | 12 months
  Comparison of the compoite outcome (consisted of : Myocardial Infarction ,stroke, Cardiovascular death) between groups

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece

REFERENCES:
- [Result] Karp A, Jacobs M, Barris B, Labkowsky A, Frishman WH. Lipoprotein(a): A Review of Risk Factors, Measurements, and Novel Treatment Modalities. Cardiol Rev. 2025 Jul-Aug 01;33(4):352-358. doi: 10.1097/CRD.0000000000000667. Epub 2024 Feb 28. PMID 38415744
- [Result] Tsimikas S, Marcovina SM. Ancestry, Lipoprotein(a), and Cardiovascular Risk Thresholds: JACC Review Topic of the Week. J Am Coll Cardiol. 2022 Aug 30;80(9):934-946. doi: 10.1016/j.jacc.2022.06.019. PMID 36007992
- [Result] Simantiris S, Antonopoulos AS, Papastamos C, Benetos G, Koumallos N, Tsioufis K, Tousoulis D. Lipoprotein(a) and inflammation- pathophysiological links and clinical implications for cardiovascular disease. J Clin Lipidol. 2023 Jan-Feb;17(1):55-63. doi: 10.1016/j.jacl.2022.10.004. Epub 2022 Oct 20. PMID 36333256
- [Result] Clarke R, Wright N, Lin K, Yu C, Walters RG, Lv J, Hill M, Kartsonaki C, Millwood IY, Bennett DA, Avery D, Yang L, Chen Y, Du H, Sherliker P, Yang X, Sun D, Li L, Qu C, Marcovina S, Collins R, Chen Z, Parish S; China Kadoorie Biobank Collaborative Group. Causal Relevance of Lp(a) for Coronary Heart Disease and Stroke Types in East Asian and European Ancestry Populations: A Mendelian Randomization Study. Circulation. 2025 Jun 17;151(24):1699-1711. doi: 10.1161/CIRCULATIONAHA.124.072086. Epub 2025 Apr 29. PMID 40297899
- [Result] Burgess S, Ference BA, Staley JR, Freitag DF, Mason AM, Nielsen SF, Willeit P, Young R, Surendran P, Karthikeyan S, Bolton TR, Peters JE, Kamstrup PR, Tybjaerg-Hansen A, Benn M, Langsted A, Schnohr P, Vedel-Krogh S, Kobylecki CJ, Ford I, Packard C, Trompet S, Jukema JW, Sattar N, Di Angelantonio E, Saleheen D, Howson JMM, Nordestgaard BG, Butterworth AS, Danesh J; European Prospective Investigation Into Cancer and Nutrition-Cardiovascular Disease (EPIC-CVD) Consortium. Association of LPA Variants With Risk of Coronary Disease and the Implications for Lipoprotein(a)-Lowering Therapies: A Mendelian Randomization Analysis. JAMA Cardiol. 2018 Jul 1;3(7):619-627. doi: 10.1001/jamacardio.2018.1470. PMID 29926099
- [Result] Larsson SC, Gill D, Mason AM, Jiang T, Back M, Butterworth AS, Burgess S. Lipoprotein(a) in Alzheimer, Atherosclerotic, Cerebrovascular, Thrombotic, and Valvular Disease: Mendelian Randomization Investigation. Circulation. 2020 Jun 2;141(22):1826-1828. doi: 10.1161/CIRCULATIONAHA.120.045826. Epub 2020 Jun 1. No abstract available. PMID 32479194
- [Result] Tsimikas S, Karwatowska-Prokopczuk E, Xia S. Lipoprotein(a) Reduction in Persons with Cardiovascular Disease. Reply. N Engl J Med. 2020 May 21;382(21):e65. doi: 10.1056/NEJMc2004861. No abstract available. PMID 32433854
- [Result] Laurent S, Cockcroft J, Van Bortel L, Boutouyrie P, Giannattasio C, Hayoz D, Pannier B, Vlachopoulos C, Wilkinson I, Struijker-Boudier H; European Network for Non-invasive Investigation of Large Arteries. Expert consensus document on arterial stiffness: methodological issues and clinical applications. Eur Heart J. 2006 Nov;27(21):2588-605. doi: 10.1093/eurheartj/ehl254. Epub 2006 Sep 25. PMID 17000623
- [Result] Lekakis J, Abraham P, Balbarini A, Blann A, Boulanger CM, Cockcroft J, Cosentino F, Deanfield J, Gallino A, Ikonomidis I, Kremastinos D, Landmesser U, Protogerou A, Stefanadis C, Tousoulis D, Vassalli G, Vink H, Werner N, Wilkinson I, Vlachopoulos C. Methods for evaluating endothelial function: a position statement from the European Society of Cardiology Working Group on Peripheral Circulation. Eur J Cardiovasc Prev Rehabil. 2011 Dec;18(6):775-89. doi: 10.1177/1741826711398179. PMID 21450600
- [Result] Paraskevaidis IA, Panou F, Papadopoulos C, Farmakis D, Parissis J, Ikonomidis I, Rigopoulos A, Iliodromitis EK, Th Kremastinos D. Evaluation of left atrial longitudinal function in patients with hypertrophic cardiomyopathy: a tissue Doppler imaging and two-dimensional strain study. Heart. 2009 Mar;95(6):483-9. doi: 10.1136/hrt.2008.146548. Epub 2008 Sep 2. PMID 18765436